CLINICAL TRIAL: NCT00396721
Title: Pilot Trial of Treatment of Poor-Prognosis IgA Nephropathy With Low Exposure to Sirolimus.
Brief Title: Sirolimus Therapy for Poor Prognosis Immunoglobulin A Nephropathy
Acronym: SIREPNA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Josep m Cruzado (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Josep m Cruzado, Nephrologist, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIREPNA/05; 2005-002610-37
Record Dates: First submitted 2006-11-03; First posted 2006-11-07 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Glomerulonephritis, IGA; Nephropathy, IGA; IGA Nephropathy
Keywords: Nephropathy, IGA; Pilot trial; Sirolimus; Rapamune
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Angiotensin-Converting Enzyme Inhibitors; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: ACE inhibitor + statin
- B (Experimental)
  Interventions: Drug: Sirolimus (study drug)+ACE inhibitor + statin

INTERVENTIONS:
Drug: ACE inhibitor + statin — sirolimus starting at 1 mg/d (target 3-6 ng/ml) plus enalapril starting at 5 mg/d to control blood pressure plus atorvastatin starting at 10 mg/d
  Arms: A
Drug: Sirolimus (study drug)+ACE inhibitor + statin — enalapril starting at 5 mg/d in order to control blood pressure. Atorvastatin starting at 10 mg/d
  Arms: B

SUMMARY:
The purpose of this study is to test in a pilot trial the efficacy and tolerance of sirolimus oral (at low doses) in patient to treat poor-prognosis IgA Nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 and with capacity to grant informed consent
* Biopsy-proven IgA nephropathy by means of standard immunohistochemical and morphological criteria
* Renal biopsy in the in the 3 months prior to randomization date
* Absence of known hepatic, cardiac, pulmonary or intestinal disease
* Glomerular filtrate estimated by Cockcroft-Gault, more than 30 ml/min
* Any of the following clinical states: a) High blood pressure defined as systolic blood pressure higher than 140 mmHg or diastolic blood pressure higher than 90 mmHg associated with proteinuria between 0.3-1 g/day and/or microhematuria. b) Proteinuria higher than 1g/day
* Women of child-bearing age will follow a suitable contraceptive method, and a negative pregnancy test will be needed before inclusion in the study

Exclusion Criteria:

* Serology positive for HIV or hepatitis B infection (defined as positive for the HbsAg antigen) or hepatitis C infection (defined as viral RNA detection)
* Treatment with steroids or immunosuppressors in the two previous years
* Evidence of active infection at the time of inclusion in the study
* Pregnancy or breastfeeding at the time of inclusion in the study
* Estimated glomerular filtration < 30 ml/min, bilirubin > 2 mg/dl, or ALT or AST two times higher than the normal upper limit
* Diabetes Mellitus, defined as patients treated with insulin or oral antidiabetics or glycemias higher than 140 mg/dl in two or more episodes
* Poor control of high blood pressure (defined as systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg, taking 3 or more antihypertensives) or evidence or suspicion of renovascular disease
* Thrombocytopenia less than 100,000 /mm3 or total neutrophil value lower than 2000 /mm3 or triglycerides value > 400 mg/dL (4.6 mmol/L) or cholesterol > 300 mg/dL (7.8 mmol/L) or LDL > 200 mg/dL
* IgA nephropathy systemic forms, i.e., Schönlein-Henoch purpura, IgA nephropathy secondary forms, post-renal transplant IgA nephropathy recurrences, cases presented in the form of rapidly progressive renal failure and cases with the presence of cellular crescents in more than 50% of the glomeruli will be excluded
* History of cancer in the previous 5 years,exception of skin basocellular carcinoma and uterine in situ carcinoma (completely removed both of them)
* Know intolerance to Sirolimus or macrolides

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-01; Primary Completion 2009-10 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of the administration of Rapamune on a clinical composite variable (change in proteinuria, blood pressure and hematuria) in patients with IgA nephropathy with poor prognosis criteria | at month 12th

SECONDARY OUTCOMES:
Change in the glomerular filtrate rate evaluated by means of radionuclide techniques (51Cr-EDTA) and comparison between both arms | At months 6th and 12th
Change in renal histology | At 12 months
Percentage of patients who withdraw from the study medication due to adverse events | Within 1 year
Percentage of patients with therapeutic failure | Within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Cruzado, Medical Doctor, Study Chair — Nephrlogy Department. Hospital Universitari de Bellvitge; Meritxell Ibernon, MD, Principal Investigator — Germans Trias i Pujol Hospital; JORDI BALLARÍN, MD, Principal Investigator — FUNDACIÓ PUIGVERT DE BARCELONA
Locations (1):
- Nephrology Department. Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Donadio JV, Grande JP. IgA nephropathy. N Engl J Med. 2002 Sep 5;347(10):738-48. doi: 10.1056/NEJMra020109. No abstract available. PMID 12213946
- [Background] Donadio JV Jr, Bergstralh EJ, Offord KP, Spencer DC, Holley KE. A controlled trial of fish oil in IgA nephropathy. Mayo Nephrology Collaborative Group. N Engl J Med. 1994 Nov 3;331(18):1194-9. doi: 10.1056/NEJM199411033311804. PMID 7935657
- [Background] Wu H, Clarkson AR, Knight JF. Restricted gammadelta T-cell receptor repertoire in IgA nephropathy renal biopsies. Kidney Int. 2001 Oct;60(4):1324-31. doi: 10.1046/j.1523-1755.2001.00937.x. PMID 11576346
- [Background] Bonegio RG, Fuhro R, Wang Z, Valeri CR, Andry C, Salant DJ, Lieberthal W. Rapamycin ameliorates proteinuria-associated tubulointerstitial inflammation and fibrosis in experimental membranous nephropathy. J Am Soc Nephrol. 2005 Jul;16(7):2063-72. doi: 10.1681/ASN.2004030180. Epub 2005 May 25. PMID 15917339
- See also: This is the center in Spain for the central contact and the main location including patients. — http://www.bellvitgehospital.cat/